CLINICAL TRIAL: NCT05117411
Title: Peripapillary Vascular Density in the Pathogenesis of Pseudophakic Cystoid Edema
Brief Title: Optical Coherence Tomography Angiography and Pseudophakic Cystoid Edema
Status: Completed | Type: Observational
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Gilda Cennamo, Principal Investigator, Federico II University
Other Study IDs: 09/21
Record Dates: First submitted 2021-09-27; First posted 2021-11-11 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2021-11

CONDITIONS: Pseudophakic Cystoid Macular Edema

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients group: Subjects over 18 years that after cataract surgery, showed pseudophakic cystoid macula edema.
  Interventions: Diagnostic Test: OCTA and pseudophakin cystoid edema
- Control Group: Normal subjects over 18 years that did not show pseudophakic cystoid macula edema.
  Interventions: Diagnostic Test: OCTA and pseudophakin cystoid edema

INTERVENTIONS:
Diagnostic Test: OCTA and pseudophakin cystoid edema — Patients underwent OCT angiografia after cataract surgery

SUMMARY:
This study evaluates the retinal vascular features in macula and papillary regions in patients affected by pseudophakic cystoid edema using optical coherence tomography angiography

DETAILED DESCRIPTION:
Pseudophakic cystoid edema represents one of the most common causes of poor visual outcome following cataratta surgery.

It is still source of debate the pathogenesis of Pseudophakic cystoid edema. Optical coherence tomography angiography represents a novel and non-invasive diagnostic technique that allows a detailed analysis of retinal vascular features. The study evaluates retrospectively the changes in optical coherence tomography angiography parameters at baseline and after three monthly after surgery.

ELIGIBILITY:
Inclusion Criteria:

* age older than 60 years
* diagnosis of pseudophakic cystoid macular oedema
* treatment-naïve for pseudophakic cystoid macular oedema
* absence of other ocular diseases, responsible for macular edema (retinal vein occlusion, diabetic retinopathy, age-related macular degeneration)

Exclusion Criteria:

* age younger than 60 years
* No diagnosis of pseudophakic cystoid macular oedema
* previous treatment for pseudophakic cystoid macular oedema
* presence of other ocular diseases, responsible for macular edema (retinal vein occlusion, diabetic retinopathy, age-related macular degeneration)

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The participans were older than 18 years with diagnosis of pseudophakic cystoid macular oedema. The participans did not present other ophthalmological diseases.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
OCTA and pseudophakic cystoid macular oedema | 3 months
  The parameters analyzed by OCTA three months after surgery are:
  Vessel density (%) of superficial capillary plexus, deep capillary plexus, coriocapillary plexus in macular region Vessel density (%) of radial peripapillary capillary plexus in papilllary region

CONTACTS AND LOCATIONS:
Overall Officials: Gilda Cennamo, Principal Investigator — Università Federico II